CLINICAL TRIAL: NCT05325619
Title: City-hospital Network: Evaluation of the Rate of Consultations in Gynecological Emergencies Under Non-emergency Management
Brief Title: Evaluation of the Rate of Consultations in Gynecological Emergencies Under "Non-urgent" Management
Acronym: URGO_CARE
Status: Completed | Type: Observational
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Other Study IDs: URGO_CARE
Record Dates: First submitted 2022-03-31; First posted 2022-04-13 (Actual); Last update posted 2023-03-07 (Actual); Status verified 2023-03

CONDITIONS: Gynecologic Disease
MeSH Terms: conditions — Genital Diseases, Female

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The difference between the demand and the current medical supply poses a real public health problem in terms of the organization of health care systems.

For several years in France, there has been an increase in the number of consultations in emergency services, particularly gynaecological ones. The two causes put forward are a change in user behavior with an increase in requests for rapid but "non-urgent" care and the inadequacy of the supply of care in the private sector.

Few studies have been carried out concerning gynaecological emergencies, unlike general emergencies.

The aim of this study is to measure the frequency of consultations in gynaecological emergencies for non-emergency reasons.

The interest of this study is therefore mainly on the optimization of the care system with the emphasis on the city-hospital network in the management of these patients.

ELIGIBILITY:
Inclusion Criteria:

* Patient whose age is ≥ 18 years
* Patient not pregnant or pregnant < 14 SA
* Patient admitted for gynecological emergency care at Paris Saint-Joseph Hospital between 01/02/2021 and 30/04/2021
* French-speaking patient

Exclusion Criteria:

* Patient under guardianship or curatorship
* Patient deprived of liberty
* Patient under court protection
* Patient objecting to the use of her data for this research

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Non-pregnant or pregnant patients < 14 weeks' gestation, admitted to the gynecological emergency department of the Paris Saint-Joseph Hospital between 01/02/2021 and 30/04/2021
Sampling Method: Non-Probability Sample
Enrollment: 809 (Actual)
Dates: Start 2022-03-23 (Actual); Primary Completion 2022-07-24 (Actual); Study Completion 2022-08-02 (Actual)

PRIMARY OUTCOMES:
Rate of gynecological emergency room visits for non-urgent reasons | Month 2
  This outcome corresponds to number of non-emergency gynecological emergency visits out of the total number of gynecological emergencies.

SECONDARY OUTCOMES:
Optimization of patient care not requiring urgent care | Month 2
  This outcome corresponds to the the number of patients who were referred to semi-emergency or semi-programmed care facilities.
Hospitalization rate | Month 2
  This outcome corresponds to the number of women hospitalized.
Surgical management rate | Month 2
  This outcome corresponds to the number of women who are operated.

CONTACTS AND LOCATIONS:
Overall Officials: Marie Charlotte Marie Charlotte, MD, Principal Investigator — Fondation Hôpital Saint-Joseph
Locations (1):
- Groupe Hospitalier Paris Saint-Joseph, Paris, France

REFERENCES:
- See also: Related Info — https://www.fncgm.com/qui-sommes-nous/la-gynecologie-medicale.html
- See also: Related Info — https://www.has-sante.fr/upload/docs/application/pdf/2017-05/dir19/urgences_soins_non_programmes_-_guide_ev_v2014.pdf
- See also: Related Info — https://www.senat.fr/rap/r16-685/r16-6852.html
- See also: Related Info — https://www.em-consulte.com/article/1094989/urgences-gynecologiques%C2%A0-etude-prospective-sur-les